### **SAB Biotherapeutics, Inc**

#### **SAB-176-101**

### A PHASE 1, RANDOMIZED DOUBLE-BLIND, PLACEBO-CONTROLLED, SINGLE ASCENDING DOSE SAFETY, TOLERABILITY, AND PHARMACOKINETICS STUDY OF SAB-176 IN HEALTHY ADULTS

#### 17AUG2020

Table, Listing, and Figure Shells

Version 1.0

Prepared by:

PPD 3900 Paramount Parkway Morrisville, NC 27560 USA

### Document History - Changes compared to previous version of SAP Shells:

| Version | Date | Changes |
|---------|------|---------|

#### General guidance

#### **Document Headers**

The following headers will be used for all tables and figures and listings outlined in this document:

```
1 mg/kg SAB-176
10 mg/kg SAB-176
25 mg/kg SAB-176
50 mg/kg SAB-176
Pooled placebo (as applicable)
Total (as applicable)
```

For all Safety tables (from 14.3.1.1 to 14.3.6.4.2) and additional Pooled SAB-176 header will be shown as applicable.

If there are no data for the entire output, then keep all titles/footnotes and column headers, remove subgroup page header where applicable, display "No data to display" as the content of the output.

#### **Document Footnotes**

The following programming footnote will be included for all tables, listings, and figures:

<DIRECTORY PATH>PROGRAM NAME Executed: DDMONYYYY hh:mm

#### Table of Contents

| General guidance | 3 |
|---|---|
| Document Headers | 3 |
| Document Footnotes | |
| Table 14.1.1 Subject Disposition All Randomized Subjects | 6 |
| Table 14.1.2 Significant Protocol Deviations | 7 |
| Table 14.1.3 Demographics Safety Population | 8 |
| Table 14.2.5.1.1 Summary of Serum Concentrations (unit) of SAB-176 Following IV Administration by Treatment PK | |
| Population | . 10 |
| Status PK Population | 11 |
| Table 14.2.5.2.1 Summary of Serum Pharmacokinetic Parameters of SAB-176 Following IV Administration by Treatment PK | |
| Population | . 12 |
| ADA Status PK Population | . 13 |
| Table 14.2.5.3.1 Statistical Assessment of Dose Proportionality of Serum Pharmacokinetic Parameters for SAB-176 PK | |
| Population | |
| Table 14.3.1.1 Overall Summary of Adverse Events Safety Population | . 15 |
| Table 14.3.1.2 Treatment-Emergent Adverse Events Safety Population | |
| Table 14.3.1.3 Treatment-Emergent Adverse Events by Relationship to Study Drug Safety Population | |
| Table 14.3.1.4 Treatment-Emergent Adverse Events by Severity Safety Population | |
| Table 14.3.4.1.1 Summary of Actual Value and Change from Baseline in Hematology Safety Population | |
| Table 14.3.4.1.2 Shift from Baseline in Hematology Safety Population | . 21 |
| Table 14.3.4.2.1 Summary of Actual Value and Change from Baseline in Serum Chemistry Safety Population | |
| Table 14.3.4.2.2 Shift from Baseline in Serum Chemistry Safety Population | |
| Table 14.3.4.3.1 Summary of Actual Value and Change from Baseline in Urianalysis Safety Population | |
| Table 14.3.4.3.2 Shift from Baseline in Urianalysis Safety Population | |
| Table 14.3.4.4.1 Summary of Actual Value and Change from Baseline in Urine biomarkers Safety Population | |
| Table 14.3.5.1 Summary of Actual Value and Change from Baseline in Vital Signs Safety Population | |
| Table 14.3.6.1.1 Summary of Anti-IgG Antibody Tilter value Safety Population | |
| Table 14.3.6.1.2 Proportion of Subjects Positive and Negative for Anti-IgG Antibody Safety Population | |
| Table 14.3.6.2.1 Summary of Anti-SAB-176 Antibody Tilter value Safety Population | |
| Table 14.3.6.2.2 Proportion of Subjects Positive and Negative for Anti-SAB-176 Antibody Safety Population | |
| Table 14.3.6.3.1 Summary of Actual Value and Change from Baseline in Serum parameters HAI assay Safety Population | |
| Table 14.3.6.3.2 Shift from Baseline in Serum parameters HAI assay Safety Population | |
| Table 14.3.6.4.1 Summary of Actual Value and Change from Baseline in Serum parameters MN assay Safety Population | |
| Table 14.3.6.4.2 Shift from Baseline in Serum parameters MN assay Safety Population | |
| Listing 16.1.7 Randomization | |
| Listing 16.2.1 Discontinued subjects Enrolled Population | |
| Listing 16.2.2.1 Admission Criteria Deviations Safety Population | |
| Listing 16.2.2.2 Protocol Deviations | |
| Listing 16.2.3 Analysis Population | |
| Listing 16.2.4.1 Demographics Safety Population | . 37 |

### SAB Biotherapeutics, Inc SAB-176-101

| Listing 16.2.4.2 Medical History Safety Population | 38 |
|---|---|
| Listing 16.2.4.4 Prior and Concomitant Medications Safety Population | 39 |
| Listing 16.2.4.5 Medical/Surgical Treatment Procedures Safety Population | 40 |
| Listing 16.2.5.1 Study Drug Administration Safety Population | 41 |
| Listing 16.2.6.1 Individual Serum Concentration of SAB-176 Safety Population | 42 |
| Listing 16.2.6.2 Individual Serum Pharmacokinetic Parameters of SAB-176 PK Population | 43 |
| Listing 16.2.7.1 Adverse Events Safety Population | 44 |
| Listing 16.2.7.2 Treatment-Related Adverse Events Safety Analysis Set | 45 |
| Listing 14.3.2.1 Serious Adverse Events Safety Population | |
| Listing 14.3.2.2 Adverse Events Leading to Early Discontinuation Safety Population | |
| Listing 16.2.8.1 Laboratory Results - Hematology Safety Population | |
| Listing 16.2.8.2 Laboratory Results - Serum Chemistry Safety Population | |
| Listing 16.2.8.3 Laboratory Results - Urinalysis Safety Population | |
| Listing 16.2.8.4 Laboratory Results - Urine biomarkers Safety Population | |
| Listing 16.2.8.5 Laboratory Results - Other Safety Population | |
| Listing 16.2.8.6 Vital Sign Results Safety Population | |
| Listing 16.2.8.7 Electrocardiogram Results Safety Population | |
| Listing 16.2.8.8 Physical Examination Safety Population | |
| Listing 16.2.8.9 Anti-IgG Antibodies using Rheumatoid factor | |
| Listing 16.2.8.10 Anti-SAB-176 Antibody | |
| Listing 16.2.8.11 Hemagglutination Inhibition (HAI) Assay Safety Population | |
| Listing 16.2.8.12 Microneutralization (MN) Assay PD Population | |
| Figure 14.2.1.1 Mean (± SD) Serum Concentration versus Time Profiles for SAB-176 PK Population | |
| Figure 14.2.1.2 Mean (± SD) Serum Concentration versus Time Profiles for SAB-176 by ADA Status PK Population | |
| Figure 14.2.2.1 Individual Serum Concentration versus Time Profiles for SAB-176 | |
| Semilogarithmic Scale | 60 |
| Figure 14.2.3.1 Scatter Plot of Individual and mean Cmax versus Dose for SAB-176 Following IV Administration PK | |
| Population | 61 |
| Figure 14.2.3.2 Scatter Plot of Individual and mean AUCO-t versus Dose for SAB-176 Following IV Administration PK | |
| Population | 62 |
| Figure 14.2.3.3 Scatter Plot of Individual and mean AUCO-inf versus Dose for SAB-176 Following IV Administration PK | |
| Population | |
| Figure 14.2.4.1 Concentration of Anti-IgG antibodies using rheumatoid factor Safety Population | |
| Figure 14.2.5.1 Concentration of Anti-SAB-176 antibody Safety Population | |
| Figure 14.2.3.1 Mean (+/-SD) Change from Baseline in Serum Type A HAI Assay Safety Population | |
| Figure 14.2.4.1 Mean (+/-SD) Change from Baseline in Serum Type A MN Assay Safety Population | 67 |

Page 5 of 67

Table 14.1.1
Subject Disposition
All Randomized Subjects

| | 1 mg/kg<br>SAB-176 | 10 mg/kg<br>SAB-176 | 25 mg/kg<br>SAB-176 | 50 mg/kg<br>SAB-176 | Pooled<br>Placebo | Total |
|---|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total Number of Subjects | | | | | | |
| Enrolled | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Randomized | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation | | | | | | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Site terminated by sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by subject | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Analysis Populations | | | | | | |
| Safety Population[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PK Population[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to Programmer: Percentages with a frequency count of zere in the Total must be suppressed.

Note: [1] The Safety population included all subjects who are randomized and received SAB-176.

All percentages are based on all randomized subjects within each treatment and overall.

Source Data: Listing 16.2.1 and Listing 16.2.3

<sup>[2]</sup> The PK population included all subjects in the safety population who have received SAB-176 treatment and have sufficient PK concentration data to calculate reliable estimates of at least one key PK parameters ( $C_{max}$  or AUC).

Table 14.1.2
Significant Protocol Deviations
All Randomized Subjects

| | 1 mg/kg<br>SAB-176<br>(N=xxx)<br>n (%) | 10 mg/kg<br>SAB-176<br>(N=xxx)<br>n (%) | 25 mg/kg<br>SAB-176<br>(N=xxx)<br>n (%) | 50 mg/kg<br>SAB-176<br>(N=xxx)<br>n (%) | Pooled<br>Placebo<br>(N=xxx)<br>n (%) | Total<br>(N=xxx)<br>n (%) |
|---|---|---|---|---|---|---|
| Number of subjects with at least one significant protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total number of significant protocol deviation | xx | XX | XX | XX | XX | XX |
| Deviation 1 Deviation 2 | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

Note: All percentages are based on Safety population within each treatment and overall.

Table 14.1.3
Demographics
Safety Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg | Pooled | |
|---|---|---|---|---|---|---|
| | SAB-176 | SAB-176 | SAB-176 | SAB-176 | Placebo | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | · · | | · · | | · · | |
| Age (Years) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Sex, n (%) | | | | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | , | , , | , | , | , | , , |
| Race, n (%) | | | | | | |
| Black or African american | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| native | | | | | | |
| Native Hawaiian or Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pacific Islander | | | | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Multi-Racial | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Screening Weight (kg) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX • X | XX • X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Screening Height (cm) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX . X | XX.X | XX.X | XX.X | XX.X |

| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
|---|---|---|---|---|---|---|
| Screening BMI (kg/m^2) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |

Note to programmer: Include all treatment groups. Summarize subjects who report two or more races as "Multiracial". If there is no such subject, remove "Multi-racial" category. Percentages with a frequency count of zero in the Total must be suppressed

Note: All percentages are based on Safety population within each treatment and overall. Source Data: Listing 16.2.4.1

Table 14.2.5.1.1

Summary of Serum Concentrations (unit) of SAB-176 Following IV Administration by Treatment PK Population

| | Scheduled Time | Summary | 1 mg/kg<br>SAB-176 | 10 mg/kg<br>SAB-176 | 25 mg/kg<br>SAB-176 | 50 mg/kg<br>SAB-176 |
|---|---|---|---|---|---|---|
| Day | (h) | Statistics | (N=xx) | (N=XX) | (N=xx) | (N=xx) |
| 0 | Pre-dose | n | XX | XX | XX | XX |
| | | Mean | XX.X | xx.x | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | xx.x | XX.X | XX.X |
| | | Geometric Mean | xx.x | xx.x | XX.X | XX.X |
| | | Geometric CV% | xx.x | xx.x | XX.X | XX.X |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Minimum | xx.x | XX.X | XX.X | XX.X |
| | | Maximum | XX.X | XX.X | XX.X | XX.X |
| | 1h post EOI | n | XX | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Geometric Mean | | | | |
| | | Geometric CV% | | | | |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Minimum | xx.x | XX.X | XX.X | XX.X |
| | | Maximum | XX.XX | XX.X | XX.X | XX.X |

#### Note to Programmer:

1. Day includes Pre-dose, 1 h post EOI, 6 h post EOI on Day 0, Day 1 Day 2, Day 3, Day 7, Day 21, Day 42 and Day 90. Note that collections beyond Day 0 will not have a 'scheduled time'.

Note: EOI = end of infusion; SOI = start of infusion

Below the limit of quantitation (BLQ) values were set to the zero for calculation of summary statistics.

ADA Status: negative

| cheduled Time (h) Pre-dose | Summary<br>Statistics | SAB-176<br>(N=xx) | SAB-176<br>(N=xx) | SAB-176<br>(N=xx) | SAB-176 |
|---|---|---|---|---|---|
| | Statistics | (N=xx) | (N=xx) | (N=vv) | |
| Pre-dose | | | | (IV-XX) | (N=xx) |
| | n | XX | XX | XX | xx |
| | Mean | xx.x | xx.x | XX.X | XX.X |
| | SD | xx.x | XX.X | XX.X | XX.X |
| | CV% | xx.x | xx.x | XX.X | XX.X |
| | Geometric Mean | xx.x | XX.X | XX.X | XX.X |
| | Geometric CV% | xx.x | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X | XX.X |
| 1h post EOI | N | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Geometric Mean | | | | |
| | Geometric CV% | | | | |
| | Median | xx.x | XX.X | XX.X | xx.x |
| | Minimum | xx.x | XX.X | XX.X | xx.x |
| | Maximum | XX.XX | xx.x | XX.X | XX.X |
| | 1h post EOI | Mean SD CV% Geometric Mean Geometric CV% Median Minimum Maximum 1h post EOI N Mean SD CV% Geometric Mean Geometric CV% Median Minimum Maximum | Mean xx.x SD xx.x CV% xx.x Geometric Mean xx.x Median xx.x Minimum xx.x Maximum xx.x 1h post EOI N xx Mean xx.x SD xx.x CV% xx.x Geometric Mean Geometric CV% Median xx.x Minimum xx.x Maximum xx.x | Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Geometric Mean xx.x xx.x Median xx.x xx.x Minimum xx.x xx.x Maximum xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Geometric Mean Geometric CV% Median xx.x xx.x Minimum xx.x xx.x Minimum xx.x xx.x Maximum xx.xx xx.x | Mean |

#### Note to Programmer:

- 1. Day includes Pre-dose, 1 h post EOI, 6 h post EOI on Day 0, Day 1, Day 2, Day 3, Day 7, Day 21, Day 42 and Day 90. Note that collections beyond Day 0 will not have a 'scheduled time'.
- 2. ADA Status includes negative, positive and/or missing

Note: EOI = end of infusion; SOI = start of infusion

Below the limit of quantitation (BLQ) values were set to the zero for calculation of summary statistics.

Table 14.2.5.2.1

Summary of Serum Pharmacokinetic Parameters of SAB-176 Following IV Administration by Treatment PK Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg |
|-------------------|---------|----------|----------|----------|
| | SAB-176 | SAB-176 | SAB-176 | SAB-176 |
| Parameters | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Cmax (unit) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X |
| CV% | xx.x | xx.x | xx.x | XX.X |
| Geometric<br>Mean | xx.x | xx.x | xx.x | xx.x |
| Geometric CV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX.X | xx.x | xx.x | XX.X |
| tmax (unit) | | | | |
| n | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX.X | XX.X | XX.X | XX.X |

#### Note to programmer:

- 1. Additional parameters: AUCO-t (unit), AUCO-O-inf (unit), t1/2 (unit), CL (unit), and Vz(unit).
- 2. Only n, median, minimum and maximum will be presented for tmax.
- 3. Geometric means are set to missing where zero values exist.

Note: AUCs, t1/2, CL, Vz will not be reported if the number of data points used to calculate  $\lambda z$  is less than 3 (not including Cmax), or the calculated coefficient of determination (R2) value for  $\lambda z$  is < 0.800 Source Data: Listing 16.2.6.2

Table 14.2.5.2.2

Summary of Serum Pharmacokinetic Parameters of SAB-176 Following IV Administration by Treatment and ADA Status
PK Population

ADA Status: negative

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg |
|-------------------|---------|----------|----------|----------|
| | SAB-176 | SAB-176 | SAB-176 | SAB-176 |
| Parameters | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Cmax (unit) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | xx.x | xx.x | XX.X |
| Geometric<br>Mean | xx.x | xx.x | xx.x | XX.X |
| Geometric CV% | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX.X | xx.x | xx.x | XX.X |
| tmax (unit) | | | | |
| n | XX | xx | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX.X | XX.X | XX.X | XX.X |

#### Note to programmer:

- 1. Additional parameters: AUCO-t (unit), AUCO-O-inf (unit), t1/2 (unit), CL (unit), and Vz(unit).
- 2. Only n, median, minimum and maximum will be presented for tmax.
- 3. Geometric means are set to missing where zero values exist.

Note: AUCs, t1/2, CL, Vz will not be reported if the number of data points used to calculate  $\lambda z$  is less than 3 (not including Cmax), or the calculated coefficient of determination (R2) value for  $\lambda z$  is < 0.800 Source Data: Listing 16.2.6.2

Table 14.2.5.3.1
Statistical Assessment of Dose Proportionality of Serum Pharmacokinetic Parameters for SAB-176
PK Population

| Dose Range | Parameter (units) | Intercept<br>Estimate | Slope<br>Estimate | Standard Error of<br>Slope | 90% CI of Slope |
|---|---|---|---|---|---|
| 1 - 50 mg/kg, IV | Cmax (unit) | X.XX | x.xx | x.xx | (x.xx, x.xx) |
| | AUC0-t(unit) | X.XX | X.XX | x.xx | (x.xx, x.xx) |
| | AUC0-inf (unit) | X.XX | X.XX | X.XX | (x.xx, x.xx) |

CI = confidence interval.

Note: Natural-log transformed pharmacokinetic parameters were analyzed using a power model where  $\ln(\text{parameter}) = \text{intercept} + \text{beta*} \ln(\text{dose})$ .

Dose proportionality is concluded if the 90% confidence interval of the slope (beta) lies entirely within (x.xxxx, x.xxxx) for dose range [i.e.  $(1+\ln(0.5)/\ln(r),1+\ln(2)/\ln(r))$ ], where r is the dose range (highest dose/lowest dose). Source Data: Listing 16.2.6.2.

Table 14.3.1.1
Overall Summary of Adverse Events
Safety Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg | Pooled | Pooled | |
|---|---|---|---|---|---|---|---|
| | SAB-176 | SAB-176 | SAB-176 | SAB-176 | SAB-176 | Placebo | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any TEAE | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Any Treatment-Related TEAE | xx | XX | XX | XX | XX | XX | XX |
| - | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| TEAE by severity | | | | | | | |
| Grade 1 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 2 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 3 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 4 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 5 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Treatment-Related TEAE by severity | | | | | | | |
| Grade 1 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 2 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 3 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 4 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Grade 5 | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Any Serious TEAE | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Any Treatment-Related Serious TEAE | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |

| Any TEAE Leading to early discontinuation | xx<br>(xx.x) | xx<br>(xx.x) | xx<br>(xx.x) | xx<br>(xx.x) | xx<br>(xx.x) | xx<br>(xx.x) | (xx.x) |
|---|---|---|---|---|---|---|---|
| Any Death | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |

Note: A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure. At each level of subject summarization, a subject is counted once if the subject reported one or more events. A treatment-related AE is defined as an AE that is evaluated by the investigator as definitely, probably, or possibly related to study drug. If the relationship information is missing, the AE will be considered related. If the severity information is missing, the AE will be considered severe. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety population within each treatment and overall.

Table 14.3.1.2
Treatment-Emergent Adverse Events
Safety Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg | Pooled | Pooled | |
|---|---|---|---|---|---|---|---|
| | SAB-176 | SAB-176 | SAB-176 | SAB-176 | SAB-176 | Placebo | Total |
| System Organ Class | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| Preferred Term | n (응) | n (%) | n (%) | n (%) | n (%) | n (응) | n (%) |
| All TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to Programmer: Include all treatment groups. System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no TEAE, then display "No treatment-emergent adverse events were reported.".

Note: A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure. At each level of subject summarization, a subject is counted once if the subject reported one or more events. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety population within each treatment and overall.

Adverse Events were coded using MedDRA, Version xx.x.

Table 14.3.1.3

Treatment-Emergent Adverse Events by Relationship to Study Drug
Safety Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg | Pooled | Pooled | |
|---|---|---|---|---|---|---|---|
| System Organ Class | SAB-176 | SAB-176 | SAB-176 | SAB-176 | SAB-176 | Placebo | Total |
| Preferred Term | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| Relationship | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| All TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unlikely Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Possibly Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Probably Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unlikely Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Possibly Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Probably Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to Programmer: Include all treatment groups. System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no TEAEs, then display "No treatment-emergent adverse events were reported.".

Note: A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure. At each level of subject summarization, a subject is counted once for the most related event. A treatment-related AE is defined as an AE that is evaluated by the investigator as definitely, probably, or possibly related to study drug. If the relationship information is missing, the AE will be considered related. In represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety population within each treatment and overall.

Adverse events were coded using MedDRA version x.x.

Table 14.3.1.4

Treatment-Emergent Adverse Events by Severity
Safety Population

| | 1 mg/kg | 10 mg/kg | 25 mg/kg | 50 mg/kg | Pooled | Pooled | |
|---|---|---|---|---|---|---|---|
| System Organ Class | SAB-176 | SAB-176 | SAB-176 | SAB-176 | SAB-176 | Placebo | Total |
| Preferred Term | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| Severity | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| All TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to Programmer: Include all treatment groups. System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no TEAEs, then display "No treatment-emergent adverse events were reported.".

Note: A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure. At each level of subject summarization, a subject is counted once if the subject reported one or more events. If the severity information is missing, the AE will be considered severe. In represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety population within each treatment and overall.

Adverse Events were coded using MedDRA, Version xx.x.

Parameter: LAB TEST #1 (UNIT)

| | | | Actua | ıl Value | | | | Chai | nge From | Baseline | [1] | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | | | | | | |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | xx.x | XX | XX | | | | | | |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | xx.x | XX | XX | | | | | | |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | | | | | | |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | | | | | | |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Day 2 | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | xx.x | XX | XX | xxx | xx.x | xx.xx | XX.X | XX | XX |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | XX.XX | xx.x | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | xx.x | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for hematology include Baseline, Day 2, Day 3, Day 7, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

# Table 14.3.4.1.2 Shift from Baseline in Hematology Safety Population

Parameter: LAB TEST #1 (UNIT)

| | | 1 m | g/kg SAB | -176 | | | Pod | oled Pla | cebo | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=xx) | | | (N=xx) | | | | |
| | | | Baseline | 9 | | | 9 | | | |
| Post-Baseline | Low | Normal | High | Total | Missing | <br>Low | Normal | High | Total | Missing |
| Visit | n (%) | n (%) | n (%) | n (%) | n | n (%) | n (%) | n (%) | n (%) | n |
| Day 2 | | | | | | | | | | |
| Low | XX | XX | XX | XX | XX | XX | XX | xx | XX | xx |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Normal | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| High | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Total | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Missing | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

...

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for hematology include Day 2, Day 3, Day 7, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

Percentages are based on the number of subjects with non-missing data at both the baseline and the corresponding post-baseline visit.

#### 

Use the same shell as Table 14.3.4.1.1.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for serum chemisty include Baseline, Day 2, Day 3, Day 7 and Day 42. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Source Data: Listing 16.2.8.2

Table 14.3.4.2.2
Shift from Baseline in Serum Chemistry
Safety Population

Use the same shell as Table 14.3.4.1.2.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for serum chemisty include Day 2, Day 3, Day 7 and Day 42. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

Percentages are based on the number of subjects with non-missing data at both the baseline and the corresponding post-baseline visit.

Table 14.3.4.3.1

Summary of Actual Value and Change from Baseline in Urianalysis

Safety Population

Use the same shell as Table 14.3.4.1.1.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for urianalysis include Baseline, Day 2, Day 3, Day 7 and Day 42. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Source Data: Listing 16.2.8.3

Table 14.3.4.3.2
Shift from Baseline in Urianalysis
Safety Population

Use the same shell as Table 14.3.4.1.2.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for urianalysis include Day 2, Day 3, Day 7 and Day 42. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

Percentages are based on the number of subjects with non-missing data at both the baseline

and the corresponding post-baseline visit.

## Table 14.3.4.4.1 Summary of Actual Value and Change from Baseline in Urine biomarkers Safety Population

Use the same shell as Table 14.3.4.1.1.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for urianalysis include Baseline, Day 2, Day 3, Day 7 and Day 42. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Table 14.3.5.1

Summary of Actual Value and Change from Baseline in Vital Signs
Safety Population

Parameter: VITAL SIGN PARAMETER #1 (UNIT)

| Visit - Time Point | | | Actua | l Value | | | | Chang | e From 1 | Baseline | [1] | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | | | | | | |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | | | | | | |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Day 1 | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | xx.x | XX | XX | XXX | XX.X | XX.XX | xx.x | XX | XX |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |

Note to Programmer: Include all treatment groups. Vital sign parameters will be displayed in the same order as the vital sign listing.

Vital Sign parameters include: systolic and diastolic blood pressure, hearth rate, respiratory rate, body temperature and pulse oximetry.

Scheduled visits for vital signs include Baseline, Day 1, Day 2, Day 3, Day 7, Day 21, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Table 14.3.6.1.1
Summary of Anti-IgG Antibody Tilter value
Safety Population

| | | | Trea | tment | |
|---|---|---|---|---|---|
| Study Day | Summary<br>Statistic | 1 mg/kg<br>SAB-176<br>(N=xx) | 10 mg/kg<br>SAB-176<br>(N=xx) | 25 mg/kg<br>SAB-176<br>(N=xx) | 50 mg/kg<br>SAB-176<br>(N=xx) |
| Predose | n | X | X | X | X |
| | Mean | XXX | XXX | XXX | XXX |
| | SD | XXX | XXX | XXX | XXX |
| | CV (%) | XXX | XXX | XXX | XXX |
| | Median | XXX | XXX | XXX | XXX |
| | Minimum | xxx | XXX | XXX | XXX |
| | Maximum | xxx | XXX | XXX | XXX |
| | Geometric Mean | XXX | XXX | XXX | XXX |
| | Geometric CV (%) | XXX | XXX | xxx | XXX |
| Day 2 | n | X | Х | x | Х |
| | Mean | XXX | XXX | XXX | XXX |
| | SD | xxx | XXX | XXX | XXX |
| | CV (%) | xxx | XXX | XXX | XXX |
| | Median | xxx | XXX | XXX | XXX |
| | Minimum | xxx | XXX | XXX | XXX |
| | Maximum | XXX | XXX | XXX | XXX |
| | Geometric Mean | xxx | XXX | XXX | XXX |
| | Geometric CV (%) | XXX | XXX | XXX | XXX |

CV = Coefficient of variation; SD = Standard deviation.

Table 14.3.6.1.2
Proportion of Subjects Positive and Negative for Anti-IgG Antibody
Safety Population

| Visit<br>Anti-IgG Antibody | 1 mg/kg<br>SAB-176<br>(N=xx) | 10 mg/kg<br>SAB-176<br>(N=xx) | 25 mg/kg<br>SAB-176<br>(N=xx) | 50 mg/kg<br>SAB-176<br>(N=xx) | Pooled SAB-<br>176<br>(N=xx) | Pooled<br>Placebo<br>(N=xx) |
|---|---|---|---|---|---|---|
| _ | | | | | | |
| Day 2 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 3 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 7 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 21 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 42 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 90 | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percentages are based on subjects within the Safety population within each treatment.

# Table 14.3.6.2.1 Summary of Anti-SAB-176 Antibody Tilter value Safety Population

Use the same shell as Table 14.3.6.1.1.

CV = Coefficient of variation; SD = Standard deviation. Source Data: Listing 16.2.8.10

Table 14.3.6.2.2

Proportion of Subjects Positive and Negative for Anti-SAB-176 Antibody
Safety Population

Use the same shell as Table 14.3.6.1.2.

Note: Percentages are based on subjects within the Safety population within each treatment.

Parameter: LAB TEST #1 (UNIT)

| | | | Actua | ıl Value | | | | Char | nge From | Baseline | [1] | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Day 7 | | | | | | | | | | | | |
| 1 mg/kg SAB-176 (N=xxx) | XXX | XX.X | xx.xx | XX.X | XX | xx | XXX | xx.x | xx.xx | XX.X | XX | XX |
| 10 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| 25 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |
| 50 mg/kg SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | XX.XX | XX.X | XX | XX |
| Pooled SAB-176 (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |
| Pooled Placebo (N=xxx) | XXX | XX.X | XX.XX | XX.X | XX | XX | XXX | XX.X | xx.xx | XX.X | XX | XX |

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for hematology include Baseline, Day 7, Day 21, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Table 14.3.6.3.2
Shift from Baseline in Serum parameters HAI assay
Safety Population

Parameter: LAB TEST #1 (UNIT)

| | | 1 m | g/kg SAB | -176 | | | Pod | oled Pla | cebo | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=xx) | | | (N=xx) | | | | |
| | | | Baseline | ) | | <br>Baseline | | | | |
| Post-Baseline | Low | Normal | High | Total | Missing | <br>Low | Normal | High | Total | Missing |
| Visit | n (%) | n (%) | n (%) | n (%) | n | n (%) | n (%) | n (%) | n (%) | n |
| Day 7 | | | | | | | | | | |
| Low | XX | XX | XX | XX | XX | XX | XX | xx | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Normal | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| High | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Total | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | | (xx.x) | (xx.x) | (xx.x) | (xx.x) | |
| Missing | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

...

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for hematology include Day 7, Day 21, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

Percentages are based on the number of subjects with non-missing data at both the baseline

and the corresponding post-baseline visit.

#### Table 14.3.6.4.1

Summary of Actual Value and Change from Baseline in Serum parameters MN assay Safety Population

Use the same shell as Table 14.3.6.3.1.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for serum chemisty include Baseline, Day 7, Day 21, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

[1] Change from baseline: post-baseline value - baseline value.

Source Data: Listing 16.2.8.12

## Table 14.3.6.4.2 Shift from Baseline in Serum parameters MN assay Safety Population

Use the same shell as Table 14.3.6.3.2.

Note to Programmer: Include all treatment groups. Lab test parameters will be displayed in the same order as the lab test listing.

Scheduled visits for serum chemisty include Day 7, Day 21, Day 42 and Day 90. Start a new page for each parameter.

Note: Baseline is defined as the last non-missing assessment prior to the study drug administration.

Percentages are based on the number of subjects with non-missing data at both the baseline and the corresponding post-baseline visit.

Listing 16.1.7 Randomization

| Subject | Cohort | Date/Time of<br>Randomization | Randomization<br>Number | Treatment |
|---|---|---|---|---|
| XXX | xxxxx | DDMMMYYYY/HH:MM | xxxxx | xxxxxxxxxxxxx |
| xxx | xxxxx | DDMMMYYYY/HH:MM | xxxxx | xxxxxxxxxxxxx |

Note to Programmer: Sort by subject and cohort.

Listing 16.2.1
Discontinued subjects
Enrolled Population

| | | | | Discontinuation | | | |
|---|---|---|---|---|---|---|---|
| Subject/<br>Cohort | Date of Last<br>Dose | Date of Final<br>Contact | Completed<br>Study? | Date | Reason | Was Blind<br>Broken? | Date/Time of<br>Unblinding |
| XXXXXXX/X | DDMMMYYYY | xxxxxx | Yes | | | No | |
| XXXXXXX/X | DDMMMYYYY | xxxxx | No | DDMMMYYYY | XXXXX | Yes | DDMMMYYYY/HH:MM |
| XXXXXXX/X | DDMMMYYYY | xxxxx | No | DDMMMYYYY | Adverse Event: XXXX | No | |

...

Note to Programmer: Sort by treatment (in the order of dose level), cohort, and subject. If discontinuation occurred due to AE, append the corresponding AE term.

## Listing 16.2.2.1 Admission Criteria Deviations Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Protocol<br>Version | Inclusion Criteria<br>Not Met | Exclusion Criteria<br>Met |
|---|---|---|---|
| XXXXXX/X | AMENDMENT X, VERSION 1.0, DD-MON-YYYY | INxx, INxx, INxx | EXxx, EXxx, EXxx |
| XXXXXX/X | AMENDMENT X, VERSION 1.0, DD-MON-YYYY | | |

Note to Programmer: Sort by treatment (in the order of dose level), cohort and subject. If there are no admission criteria deviations, then display "No admission criteria deviations were reported.".

### Listing 16.2.2.2 Protocol Deviations

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Date (Day) [1]<br>of Deviation | Important<br>Deviation | Description |
|---|---|---|---|
| XXXXXX/X | DDMMMYYYY (xx) | Yes | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX/X | DDMMMYYYY (xx) | No | XXXXXXXXXXXX |
| Note to programme | . Cout by tweetmant (in the | | cohort and subject Start a new name for each |

Note to programmer: Sort by treatment (in the order of dose level), cohort and subject. Start a new page for each treatment. If there are no protocol deviations, then display "No protocol deviations were reported."

<sup>[1]</sup> Day is calculated relative to the first dose date

### Listing 16.2.3 Analysis Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Safety Population [1] | Reason for Exclusion | PK Population [2] | Reason for Exclusion |
|---|---|---|---|---|
| XXXXXX/X | Yes | | Yes | |
| XXXXXX/X | No | xxxxxxxx | No | XXXXXXXX |

Note to programmer: Sort by treatment (in the order of dose level), cohort and subject. Start a new page for each treatment.

<sup>[1]</sup> The Safety population included all subjects who are randomized and received SAB-176.

<sup>[2]</sup> The PK population included all subjects in the safety population who have received SAB-176 treatment and have sufficient PK concentration data to calculate reliable estimates of at least one key PK parameters ( $C_{max}$  or AUC).
Listing 16.2.4.1
Demographics
Safety Population

Treatment: xx mg/kg xxxxxxxx

| | Date of | | | | | | | Screenin | g |
|---|---|---|---|---|---|---|---|---|---|
| Subject/<br>Cohort | Informed<br>Consent | Date of<br>Birth | Age(years) | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m2) |
| XXXXXX/X | DDMMMYYYY | DDMONYYYY | XX | Male | ***** | NOT<br>HISPANIC<br>OR LATINO | XXX.X | XXX.X | XXX.X |
| XXXXXX/X | DDMMMYYYY | DDMONYYYY | XX | Female | xxxxxxxx | HISPANIC<br>OR LATINO | XXX.X | XXX.X | XXX.X |

Note to Programmer: Sort by treatment (in the order of dose level), cohort and subject. Start a new page for each treatment.

Listing 16.2.4.2 Medical History Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Condition/Diagnosis | System Organ Class [1] /<br>Preferred Term [1] / | Start Date/Stop Date |
|---|---|---|---|
| XXXXXX/X | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/DDMONYYYY |
| | XXXXXXXX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/Ongoing |
| XXXXXX/X | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/DDMONYYYY |

Note to Programmer: Sort by treatment (in the order of dose level) cohort, subject, condition/diagnosis, and start/stop date. Start a new page for each treatment. Display "Ongoing" in place of Stop Date if the condition is ongoing. If there are no medical histories, then display "No medical histories were reported."

<sup>[1]</sup> From MedDRA version xx.x.

# Listing 16.2.4.4 Prior and Concomitant Medications Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Preferred Drug Name<br>[1]/<br>Drug Name | Prior to<br>Study | Individual<br>Dose/<br>Total<br>daily dose | Unit | Start Date Time (Day)/ Stop Date Time (Day) | Route/<br>Freq | Indication<br>(AE ID or MH ID) |
|---|---|---|---|---|---|---|---|
| xxxxxx/x | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YES | XXXX/<br>XXXX | XXXXXX | DDMONYYYY HH:MM (XX)/ DDMONYYYY HH:MM(XX) | XXX/XXX | XXXXXXXXX<br>(MH: XXXX) |
| XXXXXX/X | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | NO | XXXX/<br>XXX | XXXXXX | DDMONYYYY<br>HH:MM (XX)/<br>Ongoing | XXX/XXX | XXXXXXXX<br>(AE: XXXX) |

Note to Programmer: Note to Programmer: Sort by treatment, cohort, subject, preferred drug name, and date/time started. Start a new page for each treatment. Display "Ongoing" in place of Stop Date/Time if the medication is ongoing. If there are no prior or concomitant medications, then display "No prior or concomitant medications were reported.".

<sup>[1]</sup> From WHODrug version xx.x.

Day is calculated relative to the first dose date

# Listing 16.2.4.5 Medical/Surgical Treatment Procedures Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/Cohort | Treatment Procedure | Indication | AE ID | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|
| XXXXXX/X | xxxxxxxxxxxxxxxx | XXXXXXXX | XX | DDMONYYYY | DDMONYYYY | No |
| XXXXXX/X | xxxxxxxxxxxxxxxxx | ADVERSE EVENT: xx | | DDMONYYYY | DDMONYYYY | No |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, subject, procedure, and start/stop date. If procedure is ongoing then display "Ongoing" in the place of Stop Date. If the procedure was for an AE, please attach the corresponding AE ID to Reason. Start a new page for each treatment. If there are no medical or surgical treatment procedures, then display "No medical or surgical treatment procedures were reported."

Day is calculated relative to the first dose date

# Listing 16.2.5.1 Study Drug Administration Safety Population

| Subject/<br>Cohort | Treatment | Planned<br>Timepoint | Treatment Start Date/Time (Day) | Treatment<br>End<br>Date/Time<br>(Day) | Planned<br>Dose<br>(Units) | Frequency/<br>Route | Dose<br>Adjusted/<br>Reason | Dose<br>Interrupted/<br>Duration<br>(Units) | Total<br>amount<br>(Units) | Initial<br>Infusion<br>rate | Treatment<br>Completed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/X | 1 mg/kg<br>SAB-176 | Day 1 | DDMONYYYY<br>HH:MM<br>(XX) | DDMONYYYY<br>HH:MM<br>(XX) | XX(xx) | ONCE/ INTRAVENOUS | YES/<br>XXXXXXXX | YES/<br>XXX (xx) | XXX (xx) | XX<br>(mL/kg/hr) | YES |
| XXXXXX/X | Placebo | | DDMONYYYY<br>HH:MM<br>(XX) | DDMONYYYY<br>HH:MM<br>(XX) | XX(xx) | | NO | NO | XXX (xx) | XX<br>(mL/kg/hr) | NO |

Note to Programmer: Sort by cohort, subject, Start Date and time.

Day is calculated relative to the first dose date

Listing 16.2.6.1
Individual Serum Concentration of SAB-176 Following IV Administration
Safety Population

| Treatment | Subject ID | Sex/Age/Race | Day | Scheduled<br>Timepoint | Collection<br>Date/Time | Actual<br>Time<br>(day) | Time<br>Deviation<br>(h) | SAB-176<br>Conc.<br>(unit) | Comment |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | XXX | x/xxx/xx | 0 | Pre-dose | DDMMMYYYY/HH:MM | xx.x | х | BLQ | |
| | | | Ŭ | 1 h post EOI | DDMMMYYYY/HH:MM | XX.X | X | XX.X | HEMOLYZED |
| | | | | 6 h post EOI | DDMMMYYYY/HH:MM | XX.X | X | XX.X | XXXXXXXXX |
| | | | 1 | - | DDMMMYYYY/HH:MM | xx.x | X | XX.X | |
| | | | 2 | | DDMMMYYYY/HH:MM | xx.x | Х | XX.X | |
| | | | 3 | | DDMMMYYYY/HH:MM | XX.X | X | XX.X | XXXXXXXX |
| | | | 7 | | DDMMMYYYY/HH:MM | XX.X | X | XX.X | |
| | | | 21 | | DDMMMYYYY/HH:MM | XX.X | X | XX.X | |
| | | | 42 | | DDMMMYYYY/HH:MM | XX.X | X | XX.X | |
| | | | 90 | | DDMMMYYYY/HH:MM | XX.X | X | XX.X | |
| | | | | | | | • | | |

#### Note to Programmer:

- 1. Sort by Treatment, Subject ID, Day and Scheduled time point.
- 2. Treatment includes 1 mg/kg SAB-176 IV, 10 mg/kg SAB-176 IV, 25 mg/kg SAB-176 IV and 50 mg/kg SAB-176 IV.
- 3. Time points are: Pre-dose, 1 h post EOI, 6 h post EOI on Day 0, Day 1, Day 2, Day 3, Day 7, Day 21, Day 42 and Day 90. Note that collections beyond Day 0 will not have a 'scheduled time'.

W = White, B = Black or African American, P = Native Hawaiian or other Pacific Islander, A = Asian, N = American Indian or Alaska Native, M = Multiple, O = Other.

EOI = end of infusion; SOI = start of infusion

BLQ: below the lower limit of quantitation (LLOQ); LLOQ for SAB-176 in serum is xx (units).

Source Data: CRF data and concentration data.

M = Male, F = Female.

| Treatment | Subject ID | Cmax<br>(unit) | tmax<br>(unit) | AUCO-t<br>(units) | AUCO-inf<br>(units) | Lambdaz<br>(unit) | t1/2<br>(unit) | CL<br>(unit) | Vz<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| AAAAA | XXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | XXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | ••• | | | | | ••• | | | |

#### Note to Programmer:

- 1. Please sort by Treatment and Subject ID.
- 2. Treatment includes 1 mg/kg SAB-176 IV, 10 mg/kg SAB-176 IV, 25 mg/kg SAB-176 IV and 50 mg/kg SAB-176 IV.

Source Data: Listing 16.2.6.1.

Listing 16.2.7.1
Adverse Events
Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject | TEAE | System Organ Class/<br>Preferred Term/<br>Adverse Event Term | Start Date/<br>Time (Day)/<br>Stop Date/<br>Time (Day) | Frequency/<br>Outcome/<br>Serious/<br>SAE Criteria | Severity/<br>Action/<br>Other Action | Relationship/<br>Study Disc/<br>CM/CM ID |
|---|---|---|---|---|---|---|
| XXXXXX | Yes | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMONYYYY HH:MM (XX)/ DDMONYYYY HH:MM (XX) | INTERMITTENT/ RECOVERED/ YES\ XXXXXX | MILD/<br>NOT APPLICABLE/<br>XXXXXXXX | RELATED/<br>NO/<br>YES/##, ## |
| | No | | | | | |
| | | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | DDMONYYYY<br>HH:MM (XX)/<br>Ongoing | CONTINOUS/<br>UNKNOWN/<br>NO | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXXX | XXX/<br>XXX/<br>NO |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, subject, AE Start Date/Time, and alphabetically by System Organ Class, Preferred Term, and Adverse Event Reported. Display "Ongoing" in place of Stop Date/Time if the AE is ongoing.

Day is calculated relative to the first dose date

CM=Concomitant or Additional Treatment Given?; CM ID=ID of medication/therapy taken for AE

Action=Action taken with study treatment

Relationship=Relationship to study treatment

Study Disc=Caused study discontinuation?

Adverse Events were coded using MedDRA, Version xx.x.

Repeat Listing 16.2.7.1 for the following:

#### Listing 16.2.7.2 Treatment-Related Adverse Events Safety Analysis Set

Note to Programmer: Sort by treatment (in the order of dose level), cohort, subject, AE Start Date/Time, and alphabetically by System Organ Class, Preferred Term, and Adverse Event Reported. Remove "Relationship" of Column 7

Day is calculated relative to the first dose date

CM=Concomitant or Additional Treatment Given?; CM ID=ID of medication/therapy taken for AE

Action=Action taken with study treatment

Relationship=Relationship to study treatment

Study Disc=Caused study discontinuation?

Adverse Events were coded using MedDRA, Version xx.x.

Listing 14.3.2.1 Serious Adverse Events Safety Population

Use the same shell as Listing 16.2.7.1. Omit Serious from column 5.

Day is calculated relative to the first dose date

CM=Concomitant or Additional Treatment Given?; CM ID=ID of medication/therapy taken for AE

Action=Action taken with study treatment

Relationship=Relationship to study treatment

Study Disc=Caused study discontinuation?

Adverse Events were coded using MedDRA, Version xx.x.

## Listing 14.3.2.2 Adverse Events Leading to Early Discontinuation Safety Population

Use the same shell as Listing 16.2.7.1.

Day is calculated relative to the first dose date CM=Concomitant or Additional Treatment Given?; CM ID=ID of medication/therapy taken for AE Relationship=Relationship to study treatment Study Disc=Caused study discontinuation? Adverse Events were coded using MedDRA, Version xx.x.

# Listing 16.2.8.1 Laboratory Results - Hematology Safety Population

Treatment: xx mg/kg xxxxxxx

| Subject/<br>Cohort | Visit | Collection Date<br>Time (Day) | Laboratory Test | Result | Units | Flag | Reference<br>Range Comm | ents |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/X | XXXXXXX | DDMONYYYY<br>HH:MM (XX) | xxxxxxxxxxxx | XXX.X | XXXXX | | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | H NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | L NCS | XXXX-XXXXX XXXX | XXXXX |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | | | |
| | XXXXXX | DDMONYYYY<br>HH:MM (XX) R | xxxxxxxxxxxx | XXX.X | xxxxx | L CS | XXX.X-XXX.X XXXX | XXXXX |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | H NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | L NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | | XXX.X-XXX.X | |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, and subject, Laboratory Test Collection Date/Time, Lab test. For Result and Reference Range, display the number of decimal places where applicable exactly as they are in the data.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

## Listing 16.2.8.2 Laboratory Results - Serum Chemistry Safety Population

Use the same shell as Listing 16.2.8.1.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

Listing 16.2.8.3
Laboratory Results - Urinalysis
Safety Population

Use the same shell as Listing 16.2.8.1.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

## Listing 16.2.8.4 Laboratory Results - Urine biomarkers Safety Population

Use the same shell as Listing 16.2.8.1.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

Listing 16.2.8.5
Laboratory Results - Other
Safety Population

Use the same shell as Listing 16.2.8.1.

Note to Programmer: Omit flag and reference range columns.

R = Repeat.

Day is calculated relative to the first dose date

Listing 16.2.8.6 Vital Sign Results Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Visit -<br>Timepoint | Date Time (Day) | Position | Sys BP (mmHg) | Dias<br>BP<br>(mmHg) | Heart<br>Rate<br>(bpm) | Resp<br>Rate<br>(bpm) | Temp | Pulse<br>Oximetry<br>(%) | Weight<br>(kg) | BMI<br>(kg/m^2) | Comment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/X | Screening | DDMMYYYY<br>HH:MM<br>(XX) R | SITTING | XXX | XX | XXX | XX | XXX | XXX | XXX | XXX | XXXXXXXX |
| | XXXXX | DDMMYYYY<br>HH:MM<br>(XX) | SITTING | XXX | XX | XXX | XX | XXX | XXX | XXX | | XXXXXXXX |
| | XXXXX | DDMMYYYY: HH:MM (XX) | | XXX | XX | XXX | XX | XXX | XXX | XXX | | XXXXXXXX |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, subject, and Date time. Start a new page for each treatment.

Day is calculated relative to the first dose date

Sys=Systolic, Dias=Diastolic, BP=Blood Pressure, bpm=beats per minute, Resp=Respiration, Temp=Temperature R=Repeat

# Listing 16.2.8.7 Electrocardiogram Results Safety Population

Treatment: xx mg/kg xxxxxxxx

| | | Visit/ | Heart | PR | | QRS | QΤ | QTcF | RR | Interpretation/ | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject/ | Position/ | Date Time | Rate | Interval | QRS Axis | Duration | Interval | Interval | Interval | Clinically | Abnormal |
| Cohort | Method | (Day) | (beats/min) | (msec) | (degrees) | (msec) | (msec) | (msec) | (msec) | Significant | Findings |
| xxxxxx/x | SUPINE/<br>XXXXXX | XXXX/<br>DDMONYYYY<br>HH:MM<br>(XX) R | XXX | XXX | XXX | XXX | XXX | XXX | XXX | AB; NCS | XXXXX |
| XXXXXX/X | XXXXX/<br>XXXXXXX | XXXX/<br>DDMONYYYY<br>HH:MM(XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXX | AB; CS | xxxxx |
| XXXXXX/X | XXXX/<br>XXXXXX | XXXX/<br>DDMONYYYY<br>HH:MM(XX) | xxx | XXX | XXX | XXX | XXX | XXX | XXX | NORMAL | |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, subject, and Date Time.

Day is calculated relative to the first dose date

bpm=beats per minute, Int=Interval

R=Repeat, AB=Abnormal, CS=Clinically Significant, NCS=Not clinically significant

# Listing 16.2.8.8 Physical Examination Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/<br>Cohort | Visit/<br>Exam Date (Day) | Body System | Interpretation and<br>Significance | Abnormal<br>Findings |
|---|---|---|---|---|
| XXXXXX/X | XXXX/ | SKIN | ABNORMAL, CS | XXXXXXXX |
| | DDMONYYYY (XX) | ABDOMEN | NORMAL | |

Note to Programmer: Sort by treatment, cohort, subject, date/time, and body system (in the order as they appear in CRF). Start a new page for each treatment.

Day is calculated relative to the first dose date

CS=Clinically Significant, NCS=Not clinically significant

Listing 16.2.8.9
Anti-IgG Antibodies using Rheumatoid factor
Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/ | | | Sample<br>Collection | | | |
|---|---|---|---|---|---|---|
| Cohort | ADA Status | Visit | Date (Day)/Time | ADA Result | Titer | Comment |
| xxxxx/x | Positive | Day 2 | DDMMMYYYY (xx)/HH:MM | Negative | XXXXX | |
| | | Day 3 | DDMMMYYYY (xx)/HH:MM | Negative | XXXXX | XXXXXXXXXXXXXXX |
| | | Day 7 | DDMMMYYYY (xx)/HH:MM | Positive | XXXXX | |
| | | Day 21 | DDMMMYYYY (xx)/HH:MM | Negative | XXXXX | |
| | | Day 42 | DDMMMYYYY (xx)/HH:MM | Negative | XXXXX | |
| | | Day 90 | DDMMMYYYY (xx)/HH:MM | Negative | XXXXX | |

Note: ADA = Anti-drug Antibody.

Note to programmer: Sort by Treatment, Subject, and Sample Collection Datetime. If titer is not collected, then remove titer column. If additional columns if other information is collected.

#### Listing 16.2.8.10 Anti-SAB-176 Antibody Safety Population

Treatment: xx mg/kg xxxxxxxx

| Subject/ | | | Sample<br>Collection | | | |
|---|---|---|---|---|---|---|
| Cohort | ADA Status | Visit | Date (Day)/Time | ADA Result | Titer | Comment |
| xxxxxx/x | Positive | Day 2 | DDMMMYYYY (xx)/HH:MM | Negative | | |
| | | Day 3 | DDMMMYYYY (xx)/HH:MM | Negative | | |
| | | Day 7 | DDMMMYYYY (xx)/HH:MM | Positive | | |
| | | Day 21 | DDMMMYYYY (xx)/HH:MM | Negative | | |
| | | Day 42 | DDMMMYYYY (xx)/HH:MM | Negative | | |
| | | Day 90 | DDMMMYYYY (xx)/HH:MM | Negative | | |

Note: ADA = Anti-drug Antibody.

Note to programmer: Sort by Treatment, Subject, and Sample Collection Datetime. If titer is not collected, then remove titer column. If additional columns if other information is collected.

## Listing 16.2.8.11 Hemagglutination Inhibition (HAI) Assay Safety Population

Treatment: xx mg/kg xxxxxxx

| Subject/<br>Cohort | Visit | Collection Date<br>Time (Day) | Laboratory Test | Result | Units | Flag | Reference<br>Range | Comments |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/X | xxxxxxx | DDMONYYYY<br>HH:MM (XX) | XXXXXXXXXXXXX | XXX.X | XXXXX | | XXX.X-XXX.X | |
| | | *************************************** | XXXXXXXXXXXXXX | XXX.X | XXXXX | H NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | L NCS | XXX.X-XXX.X | XXXXXXXX |
| | | | XXXXXXXXXXXXX | XXX.X | XXXXX | | | |
| | xxxxxx | DDMONYYYY<br>HH:MM (XX) R | xxxxxxxxxxxx | XXX.X | xxxxx | L CS | XXX.X-XXX.X | XXXXXXXX |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | H NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | L NCS | XXX.X-XXX.X | |
| | | | XXXXXXXXXXXXXX | XXX.X | XXXXX | | XXX.X-XXX.X | |

Note to Programmer: Sort by treatment (in the order of dose level), cohort, and subject, Laboratory Test Collection Date/Time, Lab test. For Result and Reference Range, display the number of decimal places where applicable exactly as they are in the data.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

# Listing 16.2.8.12 Microneutralization (MN) Assay PD Population

Use the same shell as Listing 16.2.8.11.

R = Repeat.

L = Low; H = High; CS = Clinically Significant; NCS = Not Clinically Significant.

Day is calculated relative to the first dose date

Figure 14.2.1.1 Mean ( $\pm$  SD) Serum Concentration versus Time Profiles for SAB-176 PK Population





Note: Time points are relative to the start of infusion. Source Data: Table 14.2.5.1.1

#### Note to programmer:

Please plot mean concentration versus nominal time and overlay 4 treatments: 1 mg/kg SAB-176, 10 mg/kg SAB-176, 25 mg/kg SAB-176 and 50 mg/kg SAB-176, display treatment labels in legend.

Figure 14.2.1.2 Mean ( $\pm$  SD) Serum Concentration versus Time Profiles for SAB-176 by ADA Status PK Population





Note: Time points are relative to the start of infusion. Source Data: Table 14.2.5.1.1

Note to programmer:

- 1. Please plot mean concentration versus nominal time and overlay 4 treatments: 1 mg/kg SAB-176, 10 mg/kg SAB-176, 25 mg/kg SAB-176 and 50 mg/kg SAB-176, display treatment labels in legend.
- 2. Please continue with ADA Status: positive and/or ADA Status: missing

 $\begin{array}{c} {\rm Figure} \ 14.2.2.1 \\ {\rm Individual} \ {\rm Serum} \ {\rm Concentration} \ {\rm versus} \ {\rm Time} \ {\rm Profiles} \ {\rm for} \ {\rm SAB-176} \\ {\rm Safety} \ {\rm Population} \end{array}$ 

Treatment: XXXXX Subject ID: xxx ADA Status: xxx

Linear Scale

Actual Time (h)

Semilogarithmic Scale



Note: Time points are relative to the start of infusion. Source Data: Listing 16.2.6.1

#### Note to Programmer:

- 1. Please plot individual concentration versus actual time.
- 2. Present one subject for each plot.
- 3. Treatment includes 1 mg/kg SAB-176, 10 mg/kg SAB-176, 25 mg/kg SAB-176 and 50 mg/kg SAB-176.

Figure 14.2.3.1

Scatter Plot of Individual and mean Cmax versus Dose for SAB-176 Following IV

Administration

PK Population



Note: open symbols represent individual data and closed symbols represent mean data.

Source Data: Listing 16.2.6.2 and Table 14.2.5.2.2

Note to Programmer: Use linear scale for both X-axis and Y-axis.



Note: open symbols represent individual data and closed symbols represent mean data.

Source Data: Listing 16.2.6.2 and Table 14.2.5.2.2

Note to Programmer: Use linear scale for both X-axis and Y-axis.

Figure 14.2.3.3

Scatter Plot of Individual and mean AUCO-inf versus Dose for SAB-176 Following IV

Administration

PK Population



Note: open symbols represent individual data and closed symbols represent mean data.

Source Data: Listing 16.2.6.2 and Table 14.2.5.2.2

Note to Programmer: Use linear scale for both X-axis and Y-axis.

Figure 14.2.4.1
Concentration of Anti-IgG antibodies using rheumatoid factor Safety Population





Note: Time points are relative to the start of infusion. Source Data: Table 14.3.6.1.1

#### Note to programmer:

Please plot mean concentration versus nominal time and overlay 4 treatments: 1 mg/kg SAB-176, 10 mg/kg SAB-176, 25 mg/kg SAB-176 and 50 mg/kg SAB-176, display treatment labels in legend.







Note: Time points are relative to the start of infusion. Source Data: Table 14.3.6.2.1

Note to programmer:

Please plot mean concentration versus nominal time and overlay 4 treatments: 1 mg/kg SAB-176, 10 mg/kg SAB-176, 25 mg/kg SAB-176 and 50 mg/kg SAB-176, display treatment labels in legend.



Note to programmer: Present all treatments (exclude total) as overlay on the same plot and provide treatment labels in the legend. Continue with Serum Type B. Start a new page for each parameter. Visits include Baseline; Day 7; Day 21, Day 42 and Day 90.

Figure 14.2.4.1 Mean (+/-SD) Change from Baseline in Serum Type A MN Assay Safety Population



Note to programmer: Present all treatments (exclude total) as overlay on the same plot and provide treatment labels in the legend. Continue with Serum Type B. Start a new page for each parameter. Visits include Baseline; Day 7; Day 21, Day 42 and Day 90.